CLINICAL TRIAL: NCT04916951
Title: Oral Amoxicillin and Cephalexin Pharmacokinetics/Pharmacodynamics (PK/PD) in the Neonatal Intensive Care Unit
Brief Title: Oral Amoxicillin and Cephalexin PK/PD in Neonates
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-2877
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Infection
MeSH Terms: interventions — Amoxicillin; Cephalexin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Amoxicillin - standard-of-care dose (No Intervention): Obtain amoxicillin plasma concentrations in patients already receiving amoxicillin
- Cephalexin - standard-of-care dose (No Intervention): Obtain cephalexin plasma concentrations in patients already receiving cephalexin
- Amoxicillin - study dose (Experimental): Obtain amoxicillin plasma concentrations after a study-administered dose of amoxicillin
  Interventions: Drug: Amoxicillin
- Cephalexin - study dose (Experimental): Obtain cephalexin plasma concentrations after a study-administered dose of cephalexin
  Interventions: Drug: Cephalexin

INTERVENTIONS:
Drug: Amoxicillin — oral one-time dose of amoxicillin
  Arms: Amoxicillin - study dose
Drug: Cephalexin — oral one-time dose of cephalexin
  Arms: Cephalexin - study dose

SUMMARY:
The goal of this study is to figure out the best doses for two oral antibiotics (called amoxicillin and cephalexin) when they are used to treat infections in newborns and young infants. In order to do this, the study plans to enroll two groups of young infants who are admitted to the Children's Hospital Colorado. In the first group, infants already receiving one of these two antibiotics will be enrolled. Over a few days in the hospital, up to 5 blood samples will be collected from each infant to measure how much of the drug is in their body at different points in time after a dose. In the second group, infants who are already receiving an IV antibiotic and who are eating normally or receiving oral medications will be enrolled. These infants will receive one dose by mouth of either amoxicillin or cephalexin, in addition to the IV antibiotic already being used to treat their infection. After the oral antibiotic dose,blood will be drawn every few hours to measure how much of the drug is still in their body. Blood levels of the antibiotics will be used to calculate how much and how often both antibiotics would need to be given to treat a variety of infections that are common in infants. The study will calculate if using a single blood level can predict whether or not an infant might be at risk of the antibiotic not working well enough for them.

DETAILED DESCRIPTION:
This proposal's objective is to evaluate the pharmacokinetics and pharmacodynamics (PK/PD) of enteral amoxicillin and cephalexin in neonates and young infants admitted to the hospital, characterize age-stratified PK/PD parameters, and use these data to improve neonatal antibiotic dosing strategies. This will involve developing and validating small-volume sampling assays using dried blood spots. The study hypothesizes that there will be significant inter-individual variation in amoxicillin and cephalexin PK/PD parameters in neonates and that delayed absorption and elimination will lead to longer times to maximal concentrations (Tmax) and prolonged half-lives (T1/2), most prominently in younger ages. In addition, the study hypothesizes that high inter-individual variability will lead to unacceptably low attainment of PK/PD efficacy targets using standard dosing regimens. To address this low target attainment, the study will aim to incorporate therapeutic drug monitoring (TDM), using a serum trough concentration, into this PD model to create a method that more accurately identifies patients likely to succeed with oral (PO) dosing. Preliminary physiologically based pharmacokinetic (PBPK) modeling and intestinal transporter genotyping will also provide a foundation for future studies on the most important factors that lead to interpatient variability in PK parameters. The neonatal population has much to gain from an improved understanding of age-specific PK/PD, as well as more frequent, and earlier, intravenous (IV) to PO transition of antibiotics. The specific aims of this study are to:

Specific Aim 1: Use a population PK approach to define PK parameters of enteral amoxicillin and cephalexin in infants aged 0-60 days, stratified by age group. This will include building preliminary physiologically based pharmacokinetic (PBPK) models for each drug.

Specific Aim 2: Develop and validate amoxicillin and cephalexin dried-blood spot assays.

Specific Aim 3: Perform PD modeling 3A: Perform PD modeling (including Monte Carlo simulation) to evaluate the expected PK/PD target attainment of amoxicillin and cephalexin by age group.

3B: Identify a minimum trough threshold needed to establish 95% target attainment.

Exploratory Aim: Correlate patient genotype for H(+)/peptide transporters (PEPT) 1 and 2 and the organic-anion-transporting polypeptide (OATP) family of transporters with patient-specific PK parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Children's Hospital Colorado derived from two groups:

  * Group 1-patients specifically receiving enteral amoxicillin (with or without clavulanate) or cephalexin for any clinical indication;
  * Group 2-patients receiving any IV antibiotic who are tolerating full enteral feeds and/or enteral medications.

Exclusion Criteria:

* Across both groups, exclusion criteria are: (1) weight <2kg, (2) renal dysfunction, including the use of any renal replacement therapy, (3) significant β-lactam allergy, (4) GI disorders significantly impairing drug absorption, (5) use of external circuits that would affect the study drug's volume of distribution (e.g. ECMO), and (6) clinically significant anemia precluding study-related blood draws.

Ages: 1 Day to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Time above Minimum Inhibitory Concentration (T > MIC) | up to 24 hours
  As a surrogate of treatment efficacy for amoxicillin and cephalexin, the investigators will determine the time that free plasma concentrations (fT > MIC) of amoxicillin and cephalexin remain above the minimum inhibitory concentration (MIC) of common neonatal pathogens. Monte Carlo simulation will be used to assess for the likelihood of fT > MIC dosing goals.

SECONDARY OUTCOMES:
Clearance (CL/F) of amoxicillin and cephalexin | Plasma drug concentrations obtained within 12 hours of a dose
  In defining pharmacokinetic parameters for both amoxicillin and cephalexin, the investigators will assess the Clearance, or CL/F (L/h/kg), of both drugs.
Volume of Distribution (V/F) of amoxicillin and cephalexin | Plasma drug concentrations obtained within 12 hours of a dose
  In defining pharmacokinetic parameters for both amoxicillin and cephalexin, the investigators will assess the Volume of Distribution, or V/F (L/kg), of both drugs
Half life (T1/2) of amoxicillin and cephalexin | Plasma drug concentrations obtained within 12 hours of a dose
  In defining pharmacokinetic parameters for both amoxicillin and cephalexin, the investigators will assess the half life, or T1/2 (hours), of both drugs.
Area under the curve (AUC) of amoxicillin and cephalexin | Plasma drug concentrations obtained within 12 hours of a dose
  In defining pharmacokinetic parameters for both amoxicillin and cephalexin, the investigators will assess the area under the curve, or AUC (h*mg/L), of both drugs.
Peak serum drug concentration (Cmax) of amoxicillin and cephalexin | Plasma drug concentrations obtained within 12 hours of a dose
  In defining pharmacokinetic parameters for both amoxicillin and cephalexin, the investigators will assess the peak serum drug concentration, or Cmax (mg/L), of both drugs.
Minimum serum drug concentration (Cmin) of amoxicillin and cephalexin | Plasma drug concentrations obtained within 12 hours of a dose
  In defining pharmacokinetic parameters for both amoxicillin and cephalexin, the investigators will assess the minimum serum drug concentration, or Cmin (mg/L), of both drugs.
Time at which maximal drug concentration is achieved (Tmax) of amoxicillin and cephalexin | Plasma drug concentrations obtained within 12 hours of a dose
  In defining pharmacokinetic parameters for both amoxicillin and cephalexin, the investigators will assess the time at which maximal drug concentration is achieved, or Tmax (hours), of both drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Haynes, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No